CLINICAL TRIAL: NCT01941160
Title: A Randomized, Placebo Controlled, Parallel Group Study to Evaluate the Effect of a Probiotic Product, Lacidofil® STRONG, in Healthy Adults Taking Antibiotic Treatment
Brief Title: Effect of a Lacidofil® STRONG in Healthy Adults Taking Antibiotic Treatment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: KGK Science Inc. (Industry)
Collaborators: Lallemand Health Solutions (Industry)
Responsible Party: Principal Investigator, Dale Wilson, MD, Medical Director, KGK Science Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 13LAHL
Record Dates: First submitted 2013-08-23; First posted 2013-09-13 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-03

CONDITIONS: Antibiotic Associated Diarrhea

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Amoxicillin/Clavulanic Acid and Lacidofil® STRONG (Experimental): Participants are provided in double blinded fashion Lacidofil® STRONG to take with antibiotics
  Interventions: Dietary Supplement: Lacidofil® STRONG
- Placebo (Placebo Comparator): Participants are provided in double blinded fashion placebo to take with antibiotics
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lacidofil® STRONG — Lacidofil® STRONG capsule twice daily
  Arms: Amoxicillin/Clavulanic Acid and Lacidofil® STRONG
Dietary Supplement: Placebo — Placebo capsule twice daily
  Arms: Placebo

SUMMARY:
The objectives of this study are to evaluate stool consistency and stool frequency during and up to 8 weeks following a 7 day antibiotic treatment with Amoxicillin/Clavulanic Acid 875mg BID.

DETAILED DESCRIPTION:
It is hypothesized that the proportion of subjects having a diarrhea-like defecation, defined as a stool frequency ≥ 3 per day and/or stool consistency ≥ 5 (Bristol Stool Score) for at least 2 days will be lower in the group receiving Lacidofil® STRONG compared to the group receiving placebo and therefore mean Bristol Stool Scores will be lower in subjects receiving Lacidofil® STRONG compared to those receiving placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 to 50 years inclusive
* Body mass index 18.0 - 29.9 kg/m2
* Healthy as determined by laboratory results, medical history and physical exam
* Agrees to comply with study procedures
* Agrees not to change current dietary habits (with the exception of avoiding pro- and prebiotics) and activity/training levels during the course of the study
* Has given voluntary, written, informed consent to participate in the study

Exclusion Criteria:

* Women who are pregnant, breastfeeding, or planning to become pregnant during the course of the trial
* Body mass index ≥ 30 kg/m2
* Average number of formed bowel movements > 3 per day or < 3 per week
* Participation in a clinical research trial within 30 days prior to randomization
* Use of antibiotics within 60 days prior to randomization.
* Habitual use of pro- and/or prebiotic products. Subjects must not consume foods or supplements containing added pro- and/or prebiotics within 3 weeks prior to randomization and during the course of the study
* Use of laxatives, enemas or suppositories 1 week prior to randomization and for the duration of the study
* Follows a vegetarian or vegan diet
* Unstable medical conditions, as determined by the Qualified Investigator
* History of chronic gastrointestinal disorders including irritable bowel syndrome; chronic constipation; chronic diarrhea; dyspepsia; gastroesophageal reflux disease; diverticulitis; colitis; Crohn's disease; or any other malabsorption or gastrointestinal disorder
* Subjects with an immuno-compromised condition (e.g. AIDS, lymphoma, patients undergoing long-term corticosteroid treatment)
* Alcohol use > 2 standard alcoholic drinks per day and/or alcohol or drug abuse within past year
* Allergy or sensitivity to test product ingredients or Amoxicillin/Clavulanic Acid
* Individuals who are cognitively impaired and/or who are unable to give informed consent
* Any other condition which in the Investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2013-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
The primary outcomes are the between group difference in mean Bristol Stool Scores (consistency) and the between group difference in the mean number of bowel movements (frequency). | Up to 63 days

SECONDARY OUTCOMES:
Incidence of AAD | Up to 63 days
  Proportion of subjects having diarrhea-like defecation defined as a stool frequency ≥ 3 per a 24 h period and/or stool consistency ≥ 5 (Bristol Stool Score) for at least 2 days (48 h period)
Influence of Lacidofil® STRONG on side effects associated with antibiotic use | Up to 63 days
  Assessed by Gastrointestinal Symptom Rating Scale (GSRS) questionnaire, bowel habits, adverse effects

OTHER OUTCOMES:
Safety profile of Lacidofil® STRONG | Up to 14 days
  Assessed by measurement of biometrics, vital signs, general blood chemistry and complete blood counts

CONTACTS AND LOCATIONS:
Overall Officials: Dale Wilson, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Synergize Inc., London, Ontario, Canada